CLINICAL TRIAL: NCT00757146
Title: NICU Course and Hospital Outcome of Infants With Bronchopulmonary Dysplasia Treated Using Inhaled Nitric Oxide
Brief Title: Neonatal Intensive Care (NICU) Course and Hospital Outcome of Infants With BPD Treated Using Inhaled Nitric Oxide
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Donald Null, University of Utah / Primary Childrens Hospital
Other Study IDs: 17091
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: chronic lung disease; bronchopulmonary dysplasia; inhaled nitric oxide; premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a chart review study of neonates admitted to Primary Children's Medical Center or University of Utah NICU who had or developed a diagnosis of bronchopulmonary dysplasia (BPD) and were treated for this condition with inhaled nitric oxide (iNO) beginning after the 4th week of life. For this study BPD will be defined as need for supplemental oxygen on day 28 of life. The data collection from the medical record will gather demographics on admission (birth weight, gestational age, etc); past medical history from transferring hospitals; admission diagnoses; hospital respiratory care treatment course and laboratory/xray findings; nutrition and growth; and discharge diagnoses including all major neonatal morbidities such as absence or severity of intraventricular hemorrhage, retinopathy of prematurity, or hearing deficits. The data will be compiled and compared to data previously published on similar infants with BPD but not treated with iNO.

DETAILED DESCRIPTION:
Recent studies (e.g. Schreiber 2003)1 have prompted several large current clinical trials on the use of inhaled nitric oxide (iNO) for the prevention of bronchopulmonary dysplasia (BPD) in preterm infants. Results of these studies are not yet published and will be forthcoming Spring 2006. However, there is evidence to suggest that for patients with BPD, treatment with iNO may improve oxygenation2 and improve pulmonary blood flow by relaxing pulmonary vascular tone. 3 Also, there is a recent primate study that suggests in the face of existing BPD, treatment with iNO may decrease oxygen and ventilation requirements through a mechanism that helps preserve surfactant protein.4 Taken together, this preliminary work suggests there may be clinical benefit in treating established BPD with iNO. However, as few data exist on the clinical course of BPD patients treated with iNO, further description is necessary to evaluate iNO as a potential treatment modality for BPD. Since iNO has been used as adjunctive therapy for neonates at PCMC with serious respiratory disease, useful information on the relationship between BPD and iNO treatment may exist within our own patient population

ELIGIBILITY:
Inclusion Criteria:

* Any patient who at 28 days of life was requiring oxygen therapy in the Neonatal Intensive Care Unit and who was then treated with iNO would be eligible for chart review. Since iNO therapy has only been available for a few years, this study will attempt to capture all patients who qualify.

Exclusion Criteria:

* Any patient who received iNO treatment under an IRB study protocol after 28d of life would not be eligible for chart review.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any patient who at 28 days of life was requiring oxygen therapy in the Neonatal Intensive Care Unit and who was then treated with iNO would be eligible for chart review. Since iNO therapy has only been available for a few years, this study will attempt to capture all patients who qualify. Any patient who received iNO treatment under an IRB study protocol after 28d of life would not be eligible for chart review.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2006-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Gather descriptive information on the hospital course and outcome of infants treated with iNO who had a diagnosis of BPD. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald .Null, MD, Principal Investigator — University of Utah / Primary Childrens Hospital
Locations (1):
- Univesity of Utah / Primary Childrens Medical Center, Salt Lake City, Utah, United States